CLINICAL TRIAL: NCT00659802
Title: A Phase II, Randomized, Multi-Centre, Double-Blind, Placebo-Controlled Trial of HMPL-004 in Patients With Mild to Moderate Active Ulcerative Colitis With or Without Mesalamine
Brief Title: Phase II Study of HMPL-004 in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMPL-004-US-02
Record Dates: First submitted 2008-04-08; First posted 2008-04-16 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): Matching dose of placebo will be given orally in capsules three times per day for 56 days.
  Interventions: Drug: Placebo
- HMPL-004 low dose (Experimental): A total of 1200 mg of HMPL-004 per day in three divided doses will be given orally in capsules, 200 mg each, for 56 days.
  Interventions: Drug: HMPL-004 low dose
- HMPL-004 high dose (Experimental): A total of 1800 mg of HMPL-004 per day in three divided doses will be given orally in capsules, 200 mg each, for 56 days.
  Interventions: Drug: HMPL-004 high dose

INTERVENTIONS:
Drug: HMPL-004 low dose — HMPL-004, 400 mg (2 x 200 mg) t.i.d. (total of 1200 mg/day).
  Other Names: Chuan xinlian
  Arms: HMPL-004 low dose
Drug: Placebo — Matching dose of Placebo
  Arms: placebo
Drug: HMPL-004 high dose — HMPL-004, 600 mg (3 x 200 mg) t.i.d. (total of 1800 mg/day).
  Other Names: Chuan xinlian
  Arms: HMPL-004 high dose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HMPL-004 in patients with active mild to moderate ulcerative colitis (UC), compared with placebo.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled Phase II study conducted in North America (U.S. and Canada) and Europe (Romania and Ukraine) in patients with mild to moderate ulcerative colitis. Treatment consisted of one of 2 doses of HMPL-004 (1200 mg daily or 1800 mg daily, administered in 3 divided doses) or matching placebo. Assessment of treatment effect is based on the Mayo score. Subjects eligible for the study will include those ≥18 years of age with mild to moderate ulcerative colitis, having a Mayo score of 4 to 10, with activity confirmed by endoscopy within 2 weeks prior to study entry, and having a Mayo endoscopy score ≥1. Subjects who are using concomitant mesalamine could enter the study. The randomization will be stratified by mesalamine use or non-use.

ELIGIBILITY:
Inclusion Criteria:

* Have active confirmed mild to moderate ulcerative colitis

Exclusion Criteria:

* Diagnosed with Crohn's Disease or

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2008-02-07 (Actual); Primary Completion 2009-10-13 (Actual); Study Completion 2009-10-13 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were required to have mild to moderate ulcerative colitis to enter the study. Study was conducted at medical clinics and hospitals in the United States, Ukraine and Romania.
Groups:
- High Dose HMPL-004 (1800 mg/Day): HMPL-004 : HMPL-004, 600 mg (3 x 200 mg) t.i.d. total of 1800 mg/day.
- Low Dose HMPL-004 (1200 mg/Day): HMPL-004 : HMPL-004, 400 mg (2 x 200 mg) t.i.d. (total of 1200 mg/day).
- Placebo: Placebo, t.i.d.
Period: Overall Study
Arm/Group | High Dose HMPL-004 (1800 mg/Day) | Low Dose HMPL-004 (1200 mg/Day) | Placebo
Started | 74 | 75 (One patient was incorrectly randomized and was excluded from the efficacy analyses.) | 75
Completed | 59 | 57 | 64
Not Completed | 15 | 18 | 11

BASELINE CHARACTERISTICS:
Population: The demographic characteristics of the ITT population, all 224 subjects but 1 were included, are summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose HMPL-004 (1800 mg/Day) | Low Dose HMPL-004 (1200 mg/Day) | Placebo | Total
Number analyzed (Participants) | 74 | 74 | 75 | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.64 (13.61) | 44.3 (14.5) | 44.68 (15.21) | 44.87 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 34 | 101
  Male | 41 | 40 | 41 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Response at Week 8
Description: Clinical response at week 8, which is a decrease in the Mayo score from the baseline by ≥ 3 points AND ≥ 30% decrease in the Mayo score along with either a decrease in the rectal bleeding score ≥ 1 OR an absolute rectal bleeding score ≤ 1.
  The full Mayo Score evaluates ulcerative colitis stage, based on four parameters: stool frequency (0-3), rectal bleeding (0-3), endoscopic evaluation (0-3) and Physician's global assessment (0-3), ranging from 0 to 12. The higher score means a higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: Based on number of subjects with a non-missing value in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose HMPL-004 (1200 mg/Day) | High Dose HMPL-004 (1800 mg/Day) | Placebo
Number analyzed (Participants) | 60 | 62 | 69
Participants | 33 | 45 | 30

2. Secondary Outcome: Number of Participants With a Clinical Remission at Week 8
Description: The percentage of subjects exhibiting clinical remission (Mayo score ≤2 with no individual score >1) at week 8.
  The full Mayo Score evaluates ulcerative colitis stage, based on four parameters: stool frequency (0-3), rectal bleeding (0-3), endoscopic evaluation (0-3) and Physician's global assessment (0-3), ranging from 0 to 12. The higher score means a higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: Based on number of subjects with a non-missing value in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose HMPL-004 (1200 mg/Day) | High Dose HMPL-004 (1800 mg/Day) | Placebo
Number analyzed (Participants) | 60 | 62 | 69
Participants | 25 | 28 | 19

3. Secondary Outcome: Number of Participants With Mucosal Healing at Week 8
Description: The percentage of subjects achieving Mucosal Healing at week 8. Mucosal Healing was defined as a significant decrease from baseline in the Mayo endoscopy sub-score ≥1 and absolute score ≤1. Mayo endoscopy sub-score ranges from 0 to 12. The higher score means a higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: Based on number of subjects with a non-missing value in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose HMPL-004 (1200 mg/Day) | High Dose HMPL-004 (1800 mg/Day) | Placebo
Number analyzed (Participants) | 60 | 62 | 69
Participants | 28 | 37 | 25

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Low Dose HMPL-004 (1200 mg/Day) | High Dose HMPL-004 (1800 mg/Day) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/74 | 2/75
Other Adverse Events (participants affected / at risk) | 45/75 | 39/74 | 45/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose HMPL-004 (1200 mg/Day) (N=75) | High Dose HMPL-004 (1800 mg/Day) (N=74) | Placebo (N=75)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1
Hematocrit decreased (Investigations) | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose HMPL-004 (1200 mg/Day) (N=75) | High Dose HMPL-004 (1800 mg/Day) (N=74) | Placebo (N=75)
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 6
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Ageusia (Nervous system disorders) | 3 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 8 | 4 | 5
Migraine (Nervous system disorders) | 0 | 0 | 2
Influenza (Infections and infestations) | 2 | 2 | 4
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1
Blood glucose increased (Investigations) | 0 | 3 | 0
Blood urea increased (Investigations) | 1 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 0 | 2
Gamma-glutamyl transferase increased (Investigations) | 3 | 1 | 2
Hematocrit decreased (Investigations) | 0 | 2 | 1
Hemoglobin decreased (Investigations) | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Chest discomfort (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 2 | 0 | 3
Edema peripheral (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 3
Basophilia (Blood and lymphatic system disorders) | 0 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No